CLINICAL TRIAL: NCT01794195
Title: Role of Mesocorticolimbic Pathway in Apathy of Patients With Parkinson's Disease. - Study Using Diffusion Tensor Imaging and Fibres Tracking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-0145; 2012-A01293-40
Record Dates: First submitted 2013-02-12; First posted 2013-02-18 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson's Disease; Apathy
Keywords: Parkinson's disease; Apathy; diffusion tensor imaging; tractography
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — Diffusion Tensor Imaging

ARMS (3):
- apathetic patients with Parkinson's disease (Experimental): The objective of this study is to explore, using diffusion weighted MRI, the regions of the brain which are proposed to play a role in motivation in apathetic Parkinson's disease patients and to define more precisely the relation between dopaminergic fibres and the meso-cortico-limbic system with the help of tractography methods
  Interventions: Behavioral: Diffusion tensor imaging and fibres tracking
- non apathetic paired patients (Experimental): The objective of this study is to explore, using diffusion weighted MRI, the regions of the brain which are proposed to play a role in motivation in apathetic Parkinson's disease patients and to define more precisely the relation between dopaminergic fibres and the meso-cortico-limbic system with the help of tractography methods
  Interventions: Behavioral: Diffusion tensor imaging and fibres tracking
- healthy paired control (Experimental): The objective of this study is to explore, using diffusion weighted MRI, the regions of the brain which are proposed to play a role in motivation in apathetic Parkinson's disease patients and to define more precisely the relation between dopaminergic fibres and the meso-cortico-limbic system with the help of tractography methods
  Interventions: Behavioral: Diffusion tensor imaging and fibres tracking

INTERVENTIONS:
Behavioral: Diffusion tensor imaging and fibres tracking

SUMMARY:
Use lay language.

Apathy is one of the most under recognised, underdiagnosed and poorly managed aspects of Parkinson's disease. Depending on methodological approach of the study, its prevalence is estimated to be between 16 and 51%.

Apathy derives from a dysfunction of the dopaminergic meso cortico limbic systems, which seems to play a central role in the control of mood and motivation. The subcortical components of this system are the ventral tegmental area (VTA), the nucleus accumbens, and the constituents of the limbic system (particularly the hippocampus and amygdala), all of which are located deep inside the brain (18). The hypothesis is that depletion of striatal dopamine from regulators located in the midbrain (VTA and SNpc) in striato-thalamo-cortical circuits results in hypofunction of these circuits and the loss of frontal cortical activity, particularly within in the frontal orbital cortex, the anterior cingulate cortex and the prefrontal cortex

The objective of this study is to explore, using diffusion weighted MRI, the regions of the brain which are proposed to play a role in motivation in apathetic Parkinson's disease patients and to define more precisely the relation between dopaminergic fibres and the meso-cortico-limbic system with the help of tractography methods

DETAILED DESCRIPTION:
3 groups :

* 20 apathetic patients with Parkinson's disease
* 20 non apathetic paired patients)
* 20 healthy paired control

Description of the protocol for patients :

J0 : Inclusion visit (duration : 4h):

* motor assessment (UPDRS)
* neuropsychological and psychiatric assessment : Cognitive assessments : Mini Mental State MMS, MATTIS Apathy assessment: Apathy Inventory from Robert et al (2002); Lille apathy rating scale (LARS) ; Starkstein scale.

Depression assessment : Montgomery et Alsberg depression rating scale (MADRS)

J0+1 day : MRI (magnetic resonance imaging) acquisition (30 minutes) Multimodal MRI examinations will be performed (Diffusion-weighted data and high-resolution 3-dimensional (3D) T1- weighted as well as T2-weighted images) on each subject on a GE 3-T.

ELIGIBILITY:
Inclusion Criteria:

-

Patients :

* Men or women aged between 18 -85 years
* Patients with an idiopathic Parkinson's disease according to UKPDSBB criterias
* Non dement (MMS ≥ 26 ; MATTIS ≥ 130)
* Affiliated to National Health system
* Having given their informed consent

Healthy controls

* Men or women aged between 18 -85 years
* Affiliated to National Health system
* Having given their informed consent

Exclusion Criteria:

* Patients :
* Patients suffering of an atypical Parkinson syndrome
* Psychiatric pathology
* Severe tremor form of PD
* Depression (MADRS >16)., dementia (MMS < 26, MATTIS < 130).
* Pregnant
* Under guardianship
* In excluding period for another study
* Any contra-indication to MRI

Healthy subject

* Subject with neurological, psychiatric diseases
* Depression, dementia, apathy
* Pregnant
* Under guardianship
* In excluding period for another study
* Any contra-indication to MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy coefficient (the fractional anisotropy coefficient is computed from the eigenvalues of the diffusion tensor) | at day 1

SECONDARY OUTCOMES:
Fibres density (number of fibres / voxel) | at day 1
Bulk diffusivity index | at day 1
Apparent diffusion coefficient | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Franck DURIF, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France